CLINICAL TRIAL: NCT00575263
Title: Sodium Channel Expression in Human Teeth
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Michael Henry, Professor, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20060051H
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Dental Pulp Disease
Keywords: Pain, Sodium Channel, Dental pulp
MeSH Terms: conditions — Dental Pulp Diseases; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Extracted teeth including pulpal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Teeth: Normal molar teeth
- painful teeth: Painful molar teeth

SUMMARY:
The human tooth pulp has many nerve fibers and is a common source of pain. This study examines nerve fibers within normal and painful samples and identifies changes that can contribute to the generation of pain.

DETAILED DESCRIPTION:
The human tooth pulp is a rich source of pain fibers and is a common site of pathology that is often accompanied by spontaneous and stimulus-induced lingering pain. A common treatment modality includes the extraction of the offending tooth diagnosed with irreversible pulpitis. Extracted teeth represent an abundant source of normal and diseased human nociceptors and the evaluation of these tissues represents a powerful model to study human pain mechanisms since the character of pain, pain levels, and response to stimuli can be documented prior to extraction.

The overall objective of this study is to correlate changes in the expression of Sodium Channels (NaCh) with clinical responses to hot and cold thermal stimuli, and the expression of the associated receptors/transducers responsible for receiving that stimulus in extracted teeth with severe and spontaneous pain. Teeth requiring extraction in the clinical setting will be used for this study.

The research questions are: 1.) To evaluate quantitatively the overall NaCh and Nav 1.3, 1.6, 1.7, 1.8 1.9 isoform expressions in nerves of normal teeth as compared to diseased teeth 2.) To evaluate quantitatively hot/cold VR1 and CMR1 receptor expression in nerves of normal teeth as compared to the nerves in the modality-specific pain groups of diseased teeth 3.) To investigate the ultrastructural localization of NaCh isoforms in different fiber types and at sites that may be involved in pain generation.

ELIGIBILITY:
Inclusion Criteria:

* individuals 16-80 years old
* normal third molar(wisdom)teeth
* painful, diseased teeth requiring extraction

Exclusion Criteria:

* individuals under age 16 or above age 80
* pregnant females
* prisoners
* nonvital painful teeth

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy patients presenting to the dental clinic with an indication for extraction of their normal third molar(wisdom) teeth or diseased teeth that are associated with pain.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2006-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sodium Channel (NaCh) expression in nerves of normal teeth compared to diseased teeth. | Immediately following extration of the tooth.
  Ex vivo lab bench study utilizing extracted human teeth.

SECONDARY OUTCOMES:
Vanilloid receptor subtype-1 (VR1) and cold-and menthol-sensitive receptor-1(CMR1) expression in normal vs diseased teeth. | Immediately following extraction of tooth.
  Ex vivo bench lab study utilizing extracted human teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Henry, DDS, PhD, Principal Investigator — University of Texas Health Science Center at San Antonio, TX
Locations (1):
- University of Texas Health Science Center, San Antonio Dental School, San Antonio, Texas, United States